CLINICAL TRIAL: NCT02320305
Title: Peptide Vaccine With Glucopyranosyl Lipid A - Stable Oil-in-Water Emulsion (GLA-SE) for Patients With Resected Melanoma: A Pilot Study
Brief Title: MART-1 Antigen With or Without TLR4 Agonist GLA-SE in Treating Patients With Stage II-IV Melanoma That Has Been Removed by Surgery
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC1177; NCI-2014-02479 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1177 (Other: Mayo Clinic); P30CA015083 (NIH)
Record Dates: First submitted 2014-12-15; First posted 2014-12-19 (Estimated); Last update posted 2020-01-14 (Actual); Status verified 2019-02

CONDITIONS: Stage IIA Skin Melanoma; Stage IIB Skin Melanoma; Stage IIC Skin Melanoma; Stage IIIA Skin Melanoma; Stage IIIB Skin Melanoma; Stage IIIC Skin Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — MART-1 Antigen; glucopyranosyl lipid-A

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (MART-1 antigen and TLR4 antagonist GLA-SE) (Experimental): Patients receive MART-1 antigen and TLR4 antagonist GLA-SE IM on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: MART-1 Antigen; Drug: TLR4 Agonist GLA-SE; Other: Laboratory Biomarker Analysis
- Arm II (MART-1 antigen) (Experimental): Patients receive MART-1 antigen IM on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: MART-1 Antigen; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Biological: MART-1 Antigen — Given IM
  Other Names: Antigen LB39-AA; Antigen SK29-AA; MART-1 Tumor Antigen
Drug: TLR4 Agonist GLA-SE — Given IM
  Other Names: GLA-SE; Glucopyranosyl Lipid A in Stable Emulsion; Glucopyranosyl Lipid Adjuvant-Stable Emulsion; Toll-like Receptor 4 Agonist GLA-SE
  Arms: Arm I (MART-1 antigen and TLR4 antagonist GLA-SE)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This randomized pilot clinical trial studies melanoma antigen recognized by T-cells 1 (MART-1) antigen with or without toll-like receptor 4 (TLR4) agonist glucopyranosyl lipid A-stable oil-in-water emulsion (GLA-SE) in treating patients with stage II-IV melanoma that has been removed by surgery. Vaccines made from MART-1a peptide or antigen may help the body build an effective immune response to kill tumor cells. Giving TLR4 agonist GLA-SE with MART-1 antigen may help increase the immune response to MART-1a antigen.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the immune response of each immunization regimen to determine an optimal regimen in terms of immune response to recommend for phase II testing.

SECONDARY OBJECTIVES:

I. Evaluate the adverse events profile of each immunization regimen.

TERTIARY OBJECTIVES:

I. Describe the immunological efficacy of the vaccine preparations as measured by the frequency and interferon (IFN) gamma production of peptide-specific cytotoxic T lymphocytes (CTL).

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive MART-1 antigen and TLR4 antagonist GLA-SE intramuscularly (IM) on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive MART-1 antigen IM on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, stage II patients are followed up at 10 weeks and then at 6, 12, 18, and 24 months and stage III-IV patients are followed up at 3, 6, 9, 12, 15, 18, 21, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Central pathology review submission; Note: this review for MART-1 positivity is mandatory prior to randomization to confirm eligibility
* Human leukocyte antigen (HLA)-A2-positive
* Histologic proof of stage II, III or IV melanoma that has been completely resected or completely treated with ablative therapy (ex: stereotactic body radiosurgery, radiofrequency ablation, cryoablation) with no current evidence of disease, as demonstrated by imaging within 2 months (stage III or stage IV; must be computed tomography [CT], magnetic resonance imaging [MRI], or positron emission tomography [PET]/CT) or 6 months (stage II; may be chest x-ray, CT, MRI, or PET/CT)
* Absolute neutrophil count (ANC) >= 1500 mL
* Hemoglobin (Hgb) > 10 g/dL
* Platelets (PLT) >= 50,000 mL
* Aspartate aminotransferase (AST) =< 3 x upper limit of normal (ULN)
* Alkaline phosphatase =< 3 x ULN
* Ability to provide informed consent
* Willingness to return to Mayo Clinic Rochester for follow-up
* Life expectancy >= 12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0, 1 or 2
* For women of childbearing potential, a negative serum pregnancy test =< 7 days prior to registration
* Willingness to provide mandatory blood samples for correlative research

Exclusion Criteria:

* Uncontrolled or current infection
* Known standard therapy for the patient's disease that is potentially curative or proven capable of extending life expectancy
* Known allergy to any of the vaccine or adjuvant components, including eggs
* Any of the following prior therapies with interval since most recent treatment:

  * Chemotherapy =< 4 weeks prior to registration
  * Biologic or immunologic therapy =< 4 weeks prior to registration
  * Radiation therapy =< 4 weeks prior to registration
* Failure to fully recover from side effects of prior therapy or surgery
* Any of the following:

  * Pregnant women
  * Nursing women
  * Women of childbearing potential or their sexual partners who are unwilling to employ adequate contraception (condoms, diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.)
* Known immune deficiency, including human immunodeficiency virus (HIV) infection
* History of systemic autoimmune disease, as patients with ongoing autoimmunity may be at an increased risk of autoimmune toxicity from the study vaccine
* Current or recent (=< 4 weeks) use of immunosuppressive medications including systemic (inhaled, oral, or intravenous [IV]) corticosteroids; Note: use of corticosteroids in doses not exceeding those used for adrenal replacement is acceptable
* History of brain metastases; EXCEPTION: patients with a solitary brain metastasis that has been completely resected, and who have no ongoing central nervous system (CNS) symptoms and an MRI documenting no evidence of CNS disease at least 3 months after resection and within 30 days of registration, are eligible for treatment
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: non-melanotic skin cancer or carcinoma-in-situ of the cervix; NOTE: if there is a history of prior malignancy > 5 years prior to registration, the patient must not be receiving other cancer treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2015-12-07 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
Immune response | Up to 24 months
  A patient is considered to have achieved an immune response if there is a 2-fold or more increase from pre-treatment levels in the absolute number of vaccine peptide-specific (MART-1a-specific) CTL as measured by tetramer staining, or if the frequency of MART-1a-specific CTL is initially undetectable (< 0.05% of CD8 T cells) and becomes detectable during the vaccine treatment period. The proportion of successes will be estimated and the exact binomial 95% confidence intervals for the true immune response rate will be calculated.

SECONDARY OUTCOMES:
Adverse event rate, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 4.0 | Up to 24 months
  The maximum grade for each type of adverse event will be recorded for each patient, and frequency tables will be reviewed to determine patterns. Additionally, the relationship of the adverse event(s) to the study treatment will be taken into consideration.

OTHER OUTCOMES:
Immunological efficacy of the vaccine preparations against tumor antigen MART-1a will be described as a function of the vaccine immune adjuvant, as measured by the frequency and IFN gamma production of vaccine-peptide specific CTL | Up to 24 months
  Additional markers of immune activation will be described as a function of each vaccine preparation. Each factor will be plotted against time. Each graph will be visually inspected for trends across time. The number of patients with at least a 2-fold change in the number of cells/plasma concentration or with a level that goes from undetectable to detectable after the 1st course will be determined. The marker profile of those who derived an immune response and those who did not will be tabled to visually compare and contrast the pattern of marker-specific responses between these patient groups.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Block, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Kobayashi RH, Mandujano JF, Rehman SM, Kobayashi AL, Geng B, Atkinson TP, Melamed I, Turpel-Kantor E, Clodi E, Gupta S. Treatment of children with primary immunodeficiencies with a subcutaneous immunoglobulin 16.5% (cutaquig(R) [octanorm]). Immunotherapy. 2021 Jul;13(10):813-824. doi: 10.2217/imt-2021-0064. Epub 2021 May 6. PMID 33955240
- [Derived] Grewal EP, Erskine CL, Nevala WK, Allred JB, Strand CA, Kottschade LA, McWilliams RR, Dronca RS, Yakovich AJ, Markovic SN, Block MS. Peptide vaccine with glucopyranosyl lipid A-stable oil-in-water emulsion for patients with resected melanoma. Immunotherapy. 2020 Sep;12(13):983-995. doi: 10.2217/imt-2020-0085. Epub 2020 Aug 5. PMID 32752904